CLINICAL TRIAL: NCT06202469
Title: The Effects of 8-week Creatine Supplementation With and Without Ubiquinol on Sperm Quality Biomarkers in Normospermic and Oligospermic Men
Brief Title: Creatine and Ubiquinol for Sperm Quality
Acronym: CRESPAQ10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Principal Investigator, Sergej Ostojic, Professor, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR-24-AK15
Record Dates: First submitted 2023-12-28; First posted 2024-01-11 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Oligospermia; Sperm Count, Low
MeSH Terms: conditions — Oligospermia | interventions — TARGET 1 dietary supplement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supplement 1 (Experimental): Creatine monohydrate
  Interventions: Dietary Supplement: Supplement 1
- Supplement 2 (Experimental): Creatine monohydrate plus ubiquinol
  Interventions: Dietary Supplement: Supplement 2
- Placebo (Placebo Comparator): Inulin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement 1 — Creatine monohydrate (5 g/day)
  Arms: Supplement 1
Dietary Supplement: Supplement 2 — Creatine monohydrate (5 g/day) plus ubiquinol (200 mg/day)
  Arms: Supplement 2
Dietary Supplement: Placebo — Placebo (inulin)
  Arms: Placebo

SUMMARY:
This randomized controlled double-blind parallel-group interventional trial explores the impact of 8-week creatine supplementation, with or without ubiquinol, on sperm quality biomarkers in normospermic and oligospermic men. It aims to determine potential enhancements in sperm health to provide insights into male fertility and reproductive health improvement strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 35 years
* Sperm quality test available (at least half will have low sperm quality)
* Informed consent
* Healthy BMI (18.5 - 24.9 kg/m2)

Exclusion Criteria:

* Major chronic disease and acute injuries
* History of dietary supplement use during the past 28 days
* No consent to randomization
* Participation in other studies

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Sperm concentration | Change from baseline sperm concentration at 8 weeks
  Number of sperm per milliliter of semen

SECONDARY OUTCOMES:
Total antioxidant capacity | Change from baseline total antioxidant capacity at 8 weeks
  Level of total antioxidant capacity in semen
Creatine kinase | Change from baseline creatine kinase at 8 weeks
  Level of creatine kinase in semen
Creatine | Change from baseline creatine at 8 weeks
  Level of creatine in semen
The World Health Organisation-Five Well-Being Index (WHO-5) | Change from baseline WHO-5 at 8 weeks
  The World Health Organisation-Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing.The raw scores are transformed to a score from 0 to 100, with lower scores indicating worse well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Sergej Ostojic, MD, PhD, Principal Investigator — University of Novi Sad
Locations (1):
- FSPE Applied Bioenergetics Lab, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in sperm quality. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Only qualified researchers with academic interest in sperm quality

REFERENCES:
- [Background] Ostojic SM, Stea TH, Engeset D. Creatine as a Promising Component of Paternal Preconception Diet. Nutrients. 2022 Jan 28;14(3):586. doi: 10.3390/nu14030586. PMID 35276945
- [Derived] Nedeljkovic D, Todorovic N, Javorac D, Baltic S, Vranes M, Panic J, Kladar N, Ratgeber L, Betlehem J, Acs P, Stea TH, Engeset D, Stajer V, Ostojic SM. The effects of 8-week creatine supplementation with and without ubiquinol on sperm quality biomarkers in normospermic and oligospermic men: A randomized controlled pilot trial. Nutr Health. 2025 Oct 6:2601060251385000. doi: 10.1177/02601060251385000. Online ahead of print. PMID 41052075